CLINICAL TRIAL: NCT00807768
Title: A Phase III Trial of Pelvic Radiation Therapy Versus Vaginal Cuff Brachytherapy Followed by Paclitaxel/Carboplatin Chemotherapy in Patients With High Risk, Early Stage Endometrial Carcinoma
Brief Title: Pelvic Radiation Therapy or Vaginal Implant Radiation Therapy, Paclitaxel, and Carboplatin in Treating Patients With High-Risk Stage I or Stage II Endometrial Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0249; NCI-2009-00610 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000629591; GOG-0249 (Other: NRG Oncology); GOG-0249 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Fatigue; Neurotoxicity Syndrome; Obesity; Stage I Uterine Corpus Cancer AJCC v7; Stage II Uterine Corpus Cancer AJCC v7
MeSH Terms: conditions — Fatigue; Neurotoxicity Syndromes; Obesity | interventions — Radiotherapy, Conformal; Carboplatin; Radiotherapy, Intensity-Modulated; Brachytherapy; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (pelvic radiation therapy) (Active Comparator): Patients undergo conventional or intensity-modulated pelvic radiation therapy once daily, 5 days a week, for 5-6 weeks (total of 25-28 fractions) in the absence of disease progression or unacceptable toxicity. Patients with stage II disease or stage I disease with a confirmed diagnosis of clear cell and/or papillary serous histology may also undergo 1 or 2 intravaginal (i.e., vaginal cuff) brachytherapy boost treatments.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Radiation: Internal Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (brachytherapy, paclitaxel, carboplatin) (Experimental): Patients undergo vaginal cuff brachytherapy comprising 3-5 high-dose rate brachytherapy treatments over approximately 2 weeks or 1 or 2 low-dose rate brachytherapy treatments over 1-2 days. Beginning within 3 weeks after initiating brachytherapy, patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1. Chemotherapy repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Radiation: Internal Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo pelvic radiation therapy
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
  Arms: Arm I (pelvic radiation therapy)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II (brachytherapy, paclitaxel, carboplatin)
Radiation: Intensity-Modulated Radiation Therapy — Undergo pelvic radiation therapy
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
  Arms: Arm I (pelvic radiation therapy)
Radiation: Internal Radiation Therapy — Undergo vaginal cuff brachytherapy
  Other Names: BRACHYTHERAPY; internal radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm II (brachytherapy, paclitaxel, carboplatin)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies pelvic radiation therapy to see how well it works compared with vaginal implant radiation therapy, paclitaxel, and carboplatin in treating patients with high-risk stage I or stage II endometrial cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Implant radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether pelvic radiation therapy alone is more effective than vaginal implant radiation therapy, paclitaxel, and carboplatin in treating patients with endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if treatment with vaginal cuff brachytherapy followed by three cycles of chemotherapy reduces the rate of recurrence or death (i.e. increases recurrence-free survival) when compared to pelvic radiation therapy.

SECONDARY OBJECTIVES:

I. To compare survival between the two treatment groups. II. To compare patterns of failure between the two treatment groups. III. To compare physical functioning, fatigue and neurotoxicity between the two treatment groups.

IV. To examine associations between primary comorbid illnesses and obesity on survival, fatigue and physical functioning.

V. To evaluate the psychometric properties (such as construct validity, reliability, sensitivity to treatment and responsiveness over time) of the Patient-Reported-Outcomes Measurement Information System (PROMIS) Fatigue Short form 1, and to evaluate fatigue measurement equivalence between women with endometrial cancer and age-matched women from the general United States (US) population.

TERTIARY OBJECTIVES:

I. To evaluate the ability of gene expression signatures in early stage endometrial cancer to predict recurrence and to explore the association between gene expression signatures in early stage endometrial cancer and clinical characteristics and outcome.

II. To bank whole blood specimens for future research.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo conventional or intensity-modulated pelvic radiation therapy once daily, 5 days a week, for 5-6 weeks (total of 25-28 fractions) in the absence of disease progression or unacceptable toxicity. Patients with stage II disease or stage I disease with a confirmed diagnosis of clear cell and/or papillary serous histology may also undergo 1 or 2 intravaginal (i.e., vaginal cuff) brachytherapy boost treatments.

ARM II: Patients undergo vaginal cuff brachytherapy comprising 3-5 high-dose rate brachytherapy treatments over approximately 2 weeks or 1 or 2 low-dose rate brachytherapy treatments over 1-2 days. Beginning within 3 weeks after initiating brachytherapy, patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30-60 minutes on day 1. Chemotherapy repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* To be considered eligible to participate in this trial, all patients must have undergone hysterectomy; bilateral salpingo-oophorectomy (open or laparoscopic approach) is strongly encouraged
* Peritoneal cytology should be obtained on entering the peritoneal cavity, as described in the Gynecologic Oncology Group (GOG) Surgical Procedures Manual (https://gogmember.gog.org/manuals/pdf/surgman.pdf); pelvic and para-aortic lymphadenectomy are optional, but strongly encouraged (as staged patients enrolled on GOG-0210-molecular markers in endometrial carcinoma are eligible for this study)

  * The procedures may be performed via laparotomy or laparoscopy (including robot-assisted) as per the surgeon?s preference; the surgeon must record in the operative report whether a lymphadenectomy was performed (see link above to Surgical Procedures Manual) or not; a specific number of lymph nodes removed will not be utilized for eligibility, but the operative report should reflect that the procedure performed was consistent with the procedures described in the GOG Surgical Manual
* If either a bilateral salpingo-oophorectomy or nodal dissection was not performed, post-operative pre-treatment computed tomography (CT)/magnetic resonance imaging (MRI) is required and must not demonstrate evidence suggestive of metastatic disease (adnexa, nodes, intraperitoneal disease); post-operative, pre-treatment CT/MRI must be performed if a pelvic and para-aortic nodal dissection was not performed
* For the purposes of description, patients will be staged according to the International Federation of Gynecology and Obstetrics (FIGO) 2009 staging system; eligibility is defined based on clinical-pathologic features; patients with endometrial carcinoma (endometrioid types) confined to the corpus uteri or with endocervical glandular involvement fitting one of the following high-intermediate risk factor categories:

  * Age >= 70 years with one risk factor
  * Age >= 50 with 2 risk factors
  * Age >= 18 years with 3 risk factors
  * Risk factors: grade 2 or 3 tumor, (+) lymphovascular space invasion, outer ? myometrial invasion; patients with these risk criteria may be enrolled with either positive or negative cytology
* Patients with stage II endometrial carcinoma (any histology) with cervical stromal invasion (occult or gross involvement), with or without high-intermediate risk factors
* Patients with serous or clear cell histology (with or without other high-intermediate risk factors) are eligible provided the disease is uterine-confined (with or without cervical stromal invasion or endocervical glandular involvement), and with peritoneal cytology negative for malignancy
* Patients must have GOG performance status 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,500/mcl (equivalent to Common Toxicity Criteria [CTCAE version [v] 3.0] grade 1)
* Platelets >= 100,000/mcl (CTCAE v3.0 grade 0-1)
* Serum creatinine =< institutional upper limit normal (ULN), CTCAE v 3.0 grade 0

  * Note: If serum creatinine > ULN, a 24-hour creatinine clearance must be collected and must be > 50 mL/min
* Bilirubin =< 1.5 x ULN (CTCAE v3.0 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 x ULN (CTCAE grade 0-1)
* Alkaline phosphatase =< 2.5 x ULN (CTCAE grade 0-1)
* Neuropathy (sensory and motor) =< CTCAE v3.0 grade 1
* Patients who have met the pre-entry requirements; testing values/results must meet eligibility criteria
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients who have already received non-surgical therapy for endometrial cancer including chemotherapy, radiation (example, pre-operative or post-operative brachytherapy), hormonal or biologic therapy
* Patients identified with pathologically confirmed spread of cancer beyond the uterus and cervix to pelvic or para-aortic lymph nodes, adnexal structures, and/or other anatomic sites, or patients with serous or clear cell histology and with positive cytologic washings
* Patients with nodal (for patients who did not have nodal dissection performed) or distant disease determined based on imaging studies; patients with suspicious nodes that have been biopsied (re-staging operation, fine needle aspiration [FNA]) and are pathologically negative will be eligible
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last 5 years; patients are excluded if their previous cancer treatment contraindicates this protocol therapy; specifically, patients who have received prior radiotherapy directed to treat disease within the abdominal cavity or pelvis are excluded
* Prior radiation of localized cancer of the breast, head and neck, thyroid, or skin is permitted, provided that it was completed more than 5 years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than 5 years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have contraindications to pelvic radiation therapy (RT) (e.g. pelvic kidney, connective tissue disease, inflammatory bowel disease, etc.) should be screened in advance and not be considered eligible for the trial
* Patients with recurrent endometrial cancer
* Patients with surgical or clinical, FIGO 2009 stage III or IV endometrial carcinoma
* Patients with non-epithelial uterine malignancies such as uterine carcinosarcoma or leiomyosarcoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2009-03-23 (Actual); Primary Completion 2014-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus E Randall, Principal Investigator — NRG Oncology
Locations (540):
- United States (533):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Southeast Gynecologic Oncology Associates, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Florida Institute of Research Medicine and Surgery-Cancer Center, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Franciscan Saint Margaret Health-Dyer Campus, Dyer, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Saint Margaret Health-Hammond Campus, Hammond, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Elliot Hospital, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Saint Luke's Hospital-Warren Campus, Phillipsburg, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University Radiation Oncology, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Chattanooga Gynecological Oncology, Chattanooga, Tennessee
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Tennessee Oncology PLLC- Centennial Medical Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - The Klabzuba Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology-Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Cancer Institutes of Washington PLLC, Yakima, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- South Korea (7):
  - Inha University, Jung-gu, Incheon
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Yongdong Severence Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Randall ME, Filiaci V, McMeekin DS, von Gruenigen V, Huang H, Yashar CM, Mannel RS, Kim JW, Salani R, DiSilvestro PA, Burke JJ, Rutherford T, Spirtos NM, Terada K, Anderson PR, Brewster WR, Small W, Aghajanian CA, Miller DS. Phase III Trial: Adjuvant Pelvic Radiation Therapy Versus Vaginal Brachytherapy Plus Paclitaxel/Carboplatin in High-Intermediate and High-Risk Early Stage Endometrial Cancer. J Clin Oncol. 2019 Jul 20;37(21):1810-1818. doi: 10.1200/JCO.18.01575. Epub 2019 Apr 17. PMID 30995174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG 0249 accrued 601 patients from March 2009 to February 2013.
Period: Overall Study
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin)
Started | 301 | 300
Completed | 301 | 300
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin) | Total
Number analyzed (Participants) | 301 | 300 | 601
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 22 | 16 | 38
  50-59 years | 95 | 72 | 167
  60-69 years | 115 | 137 | 252
  >=70 years | 69 | 75 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301 | 300 | 601
  Male | 0 | 0 | 0
Cell Type [Count of Participants; unit: Participants] — Grade 1 endometrioid endometrial cancers are well differentiated. Grade 2 tumors are moderately differentiated. Grade 3 tumors are poorly differentiated. Lower grades have a higher relapse free survival rate..
  Participants
    Endometrioid, grade 1 | 50 | 56 | 106
    Endometrioid, grade 2 | 109 | 103 | 212
    Endometrioid, grade 3 or not graded | 63 | 63 | 126
    Serous | 46 | 42 | 88
    Clear Cell | 15 | 13 | 28
    Mixed | 14 | 17 | 31
    Other | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence or Death Events at Primary Analysis
Description: Recurrence-Free Survival is the period from study entry until disease recurrence, death, or date of last contact
Time Frame: Within 4 weeks after completing or discontinuing study therapy, then every 6 months for 2 years, then annually for 3 years, then as clinically indicated, assessed up to 10 years
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 301 | 300
Participants | 44 | 43

2. Secondary Outcome: Number of Participants With Death Events
Description: The number of death events is reported. Overall survival is reported by the number of deaths occurring while on study.
Time Frame: Overall survival is measured from study enrollment for up to 10 years.
Population: All enrolled patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 301 | 300
Participants | 39 | 37

3. Secondary Outcome: Number of Participants With Sites of Recurrence
Description: Three competing risk analyses were carried out for three different types of recurrences: 1) any vaginal, 2) any pelvic or any PA nodes and 3) any distant. More than one type of recurrence can be counted for an individual patient. A death prior to a specific type of recurrence was considered a competing event.
Time Frame: Within 4 weeks after completing or discontinuing study therapy, then every 6 months for 2 years, then annually for 3 years, then as clinically indicated thereafter, up to 10 years
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 301 | 300
Participants
  Vaginal recurrence | 6 | 6
  Pelvic or PA node | 12 | 25
  Distant recurrence | 47 | 47

4. Secondary Outcome: Patient Reported Fatigue
Description: Patient reported fatigue as measured with the Functional Assessment of Chronic Illness Therapy- Fatigue scale (FACIT-Fatigue). The FACIT-Fatigue contains 13 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative items, reversal was performed prior to score calculation. According to the FACIT measurement system, the Fatigue score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the scale. The FACIT-Fatigue score ranges 0-52 with a large score suggests less fatigue.
Time Frame: Prior to study treatment (baseline), 4 weeks post the starting of study treatment, 10-11 weeks post the starting of study treatment, 8 months post the starting of study treatment, 14 months post the starting of study treatment
Population: Provided baseline and >= follow-up assessments
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 263 | 277
units on a scale
  Baseline | 40.5 (0.6) | 41.2 (0.6)
  4 Weeks | 35.8 (0.7) | 35.8 (0.6)
  10-11 Weeks | 40.5 (0.6) | 36.8 (0.7)
  8 Months | 42.1 (0.5) | 40.3 (0.6)
  14 Months | 40.9 (0.6) | 41.1 (0.6)

5. Secondary Outcome: Patient-reported Neurotoxicity
Description: Patient reported neurotoxicity symptoms as measured with the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - neurotoxicity subscale (short version) (FACT/GOG-Ntx subscale). The FACT/GOG-Ntx subscale contains 4 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative items, reversal was performed prior to score calculation. According to the FACIT measurement system, the Ntx score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the scale. The Ntx score ranges 0-16 with a large score suggesting less neurotoxicity.
Time Frame: as for outcome 4
Population: Provided baseline and ≥ follow-up assessments
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 263 | 277
units on a scale
  Baseline | 14.6 (0.2) | 14.7 (0.1)
  4 Weeks | 14.6 (0.1) | 13.0 (0.2)
  10-11 Weeks | 14.2 (0.1) | 12.0 (0.2)
  8 Months | 14.0 (0.2) | 12.7 (0.2)
  14 Months | 13.5 (0.2) | 12.8 (0.2)

6. Secondary Outcome: Patient-reported Quality of Life
Description: Patient reported quality of life as measured with the Treatment Outcome Index of the Functional Assessment of Cancer Therapy for endometrial cancer (FACT-En TOI). The FACT-En TOI is a scale for assessing general QOL of endometrial cancer patients. It consists of three subscales: Physical Well Being (7 items), Functional Well Being (7 items), and Endometrium Cancer subscale (16 items). Each item in the FACT-En TOI was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). . The FACT-En TOI score is calculated as the sum of the subscale scores if more than 80% of the FACT-En TOI items provide valid answers and all of the component subscales have valid scores. The FACT-En TOI score ranges 0-120 with a large score suggests better QOL
Time Frame: as for outcome 4
Population: Provided baseline and >= follow-up assessments
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 263 | 277
units on a scale
  Baseline | 98.5 (0.9) | 98.7 (0.9)
  4 Weeks | 91.0 (0.9) | 92.2 (0.8)
  10-11 Weeks | 98.7 (0.9) | 95.6 (0.8)
  8 Months | 101.5 (0.8) | 99.9 (0.9)
  14 Months | 99.7 (1.0) | 102.1 (0.9)

7. Other Pre Specified Outcome: Gene Expression Based Risk Score
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs were assessed from the date of treatment initiation up to 30 days after the last cycle of treatment. Median treatment duration is approximately 8 weeks.
Arm/Group | Arm I (Pelvic Radiation Therapy) | Arm II (Brachytherapy, Paclitaxel, Carboplatin)
Serious Adverse Events (participants affected / at risk) | 9/283 | 32/290
Other Adverse Events (participants affected / at risk) | 245/283 | 284/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Pelvic Radiation Therapy) (N=283) | Arm II (Brachytherapy, Paclitaxel, Carboplatin) (N=290)
Neutrophils (Blood and lymphatic system disorders) | 0 | 11
Platelets (Blood and lymphatic system disorders) | 0 | 1
Leukocytes (Blood and lymphatic system disorders) | 0 | 1
Cardipulmonary Arrest (Cardiac disorders) | 1 | 0
Death No Ctcae Term - Death Nos (General disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Febrile Neutropenia (Infections and infestations) | 0 | 3
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Mood Alteration - Anxiety (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 0 | 1
Pain: Chest Wall (General disorders) | 0 | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0
Peripheral Arterial Ischemia (Vascular disorders) | 0 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Pelvic Radiation Therapy) (N=283) | Arm II (Brachytherapy, Paclitaxel, Carboplatin) (N=290)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1 | 17
Rhinitis (Immune system disorders) | 0 | 4
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 4
Neutrophils (Blood and lymphatic system disorders) | 31 | 227
Platelets (Blood and lymphatic system disorders) | 42 | 135
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 | 5
Leukocytes (Blood and lymphatic system disorders) | 107 | 234
Lymphopenia (Blood and lymphatic system disorders) | 20 | 16
Hemoglobin (Blood and lymphatic system disorders) | 93 | 206
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 7
S/N Arrhythmia: Atrial Flutter (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 0 | 2
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 0 | 2
Hypertension (Cardiac disorders) | 6 | 13
Cardiac General - Other (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 1 | 3
Inr (Vascular disorders) | 0 | 2
Coagulopathy - Other (Vascular disorders) | 0 | 1
Ptt (Vascular disorders) | 0 | 1
Sweating (General disorders) | 0 | 3
Weight Gain (General disorders) | 3 | 3
Fever (General disorders) | 2 | 3
Weight Loss (General disorders) | 6 | 6
Rigors/Chills (General disorders) | 2 | 6
Fatigue (General disorders) | 116 | 192
Insomnia (General disorders) | 11 | 32
Nail Changes (Skin and subcutaneous tissue disorders) | 0 | 5
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 3 | 188
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis - Chemoradiation (Skin and subcutaneous tissue disorders) | 0 | 1
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 2 | 0
Bruising (Skin and subcutaneous tissue disorders) | 3 | 5
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 36
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 5
Dermatitis - Radiation (Skin and subcutaneous tissue disorders) | 20 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 14
Burn (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 0 | 6
Hand-Foot (Skin and subcutaneous tissue disorders) | 0 | 3
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 4 | 6
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 4
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Hot Flashes (Endocrine disorders) | 11 | 17
Diabetes (Endocrine disorders) | 1 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 5 | 0
Proctitis (Gastrointestinal disorders) | 4 | 1
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 6 | 6
Heartburn (Gastrointestinal disorders) | 4 | 16
Mucositis (Functional/Sympt) - Larynx (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 3
Distention (Gastrointestinal disorders) | 2 | 2
Taste Alteration (Gastrointestinal disorders) | 5 | 25
Incontinence, Anal (Gastrointestinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 2
Mucositis (Functional/Sympt) - Rectum (Gastrointestinal disorders) | 1 | 0
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 1 | 13
Colitis (Gastrointestinal disorders) | 1 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 0 | 11
Vomiting (Gastrointestinal disorders) | 9 | 47
Anorexia (Gastrointestinal disorders) | 21 | 51
Dehydration (Gastrointestinal disorders) | 3 | 9
Constipation (Gastrointestinal disorders) | 27 | 102
Nausea (Gastrointestinal disorders) | 55 | 114
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 155 | 83
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 0 | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 1 | 6
Hemorrhage, Gu - Urethra (Vascular disorders) | 1 | 0
Hemorrhage, Gi - Rectum (Vascular disorders) | 3 | 6
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 0 | 5
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Anus (Vascular disorders) | 1 | 1
Petechiae (Vascular disorders) | 0 | 1
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 | 0
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Soft Tissue Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1 | 0
Febrile Neutropenia (Infections and infestations) | 0 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Lip/Perioral (Infections and infestations) | 0 | 1
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 0
Inf Unknown Anc: Sinus (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 6 | 9
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1 | 1
Infection - Other (Infections and infestations) | 4 | 3
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 0 | 2
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 0 | 1
Inf Unknown Anc: Vagina (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 0 | 2
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Paranasal (Infections and infestations) | 0 | 1
Inf Unknown Anc: Lymphatic (Infections and infestations) | 1 | 0
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 0 | 11
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 2 | 2
Inf Unknown Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Vagina (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Sinus (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 1 | 2
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 0 | 3
Lymphedema-Related Fibrosis (Blood and lymphatic system disorders) | 1 | 0
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 1 | 0
Edema: Limb (Blood and lymphatic system disorders) | 15 | 25
Edema: Head And Neck (Blood and lymphatic system disorders) | 0 | 1
Ast (Metabolism and nutrition disorders) | 1 | 9
Gfr (Metabolism and nutrition disorders) | 1 | 0
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 0 | 7
Cholesterol,serum High (Metabolism and nutrition disorders) | 0 | 2
Proteinuria (Metabolism and nutrition disorders) | 0 | 6
Hemoglobinuria (Metabolism and nutrition disorders) | 1 | 1
Creatinine (Metabolism and nutrition disorders) | 1 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 9
Ggt (Metabolism and nutrition disorders) | 0 | 1
Alt (Metabolism and nutrition disorders) | 3 | 10
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3 | 13
Bilirubin (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 12
Hyponatremia (Metabolism and nutrition disorders) | 2 | 14
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 2
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 10
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 43
Hypokalemia (Metabolism and nutrition disorders) | 4 | 23
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 30
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint-Function (Musculoskeletal and connective tissue disorders) | 0 | 1
Extremity-Upper (Function) (Musculoskeletal and connective tissue disorders) | 0 | 1
Gait/Walking (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 5 | 8
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 3 | 4
Syncope (Nervous system disorders) | 2 | 2
Involuntary Movement (Nervous system disorders) | 0 | 1
Neurology - Other (Nervous system disorders) | 1 | 0
Mood Alteration - Depression (Nervous system disorders) | 6 | 9
Mood Alteration - Anxiety (Nervous system disorders) | 7 | 16
Mood Alteration - Agitation (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 2
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Cognitive Disturbance (Nervous system disorders) | 0 | 3
Memory Impairment (Nervous system disorders) | 1 | 7
Dizziness (Nervous system disorders) | 5 | 13
Neuropathy-Sensory (Nervous system disorders) | 13 | 146
Neuropathy-Motor (Nervous system disorders) | 1 | 13
Ocular/Visual - Other (Eye disorders) | 1 | 0
Watery Eye (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Flashing Lights/Floaters (Eye disorders) | 0 | 4
Blurred Vision (Eye disorders) | 2 | 14
Pain - Other (General disorders) | 6 | 2
Pain: Urethra (General disorders) | 14 | 7
Pain: Perineum (General disorders) | 3 | 2
Pain: Pelvis (General disorders) | 9 | 7
Pain: Breast (General disorders) | 0 | 2
Pain: Vagina (General disorders) | 2 | 10
Pain: Chest /Thorax Nos (General disorders) | 0 | 2
Pain: Chest Wall (General disorders) | 0 | 3
Pain: Throat/Pharynx/Larynx (General disorders) | 0 | 1
Pain: Head/Headache (General disorders) | 6 | 34
Pain: Neck (General disorders) | 1 | 1
Pain: Intestine (General disorders) | 1 | 1
Pain: Extremity-Limb (General disorders) | 5 | 19
Pain: Back (General disorders) | 10 | 10
Pain: Joint (General disorders) | 3 | 69
Pain: Bone (General disorders) | 3 | 21
Pain: Kidney (General disorders) | 1 | 0
Pain: Bladder (General disorders) | 7 | 3
Pain: Pain Nos (General disorders) | 1 | 6
Pain: Stomach (General disorders) | 2 | 2
Pain: Rectum (General disorders) | 4 | 2
Pain: Abdominal Pain Nos (General disorders) | 34 | 24
Pain: Scalp (General disorders) | 0 | 1
Pain: Skin (General disorders) | 1 | 1
Pain: Middle Ear (General disorders) | 0 | 3
Pain: Face (General disorders) | 0 | 1
Pain: Muscle (General disorders) | 6 | 53
Pain: Anus (General disorders) | 2 | 0
Pain: Neuralgia (General disorders) | 0 | 2
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 30
Renal/Genitourinary - Other (Renal and urinary disorders) | 4 | 5
Cystitis (Renal and urinary disorders) | 13 | 6
Urinary Retention (Renal and urinary disorders) | 1 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 1
Incontinence, Urinary (Renal and urinary disorders) | 9 | 14
Bladder Spasm (Renal and urinary disorders) | 2 | 1
Urinary Frequency (Renal and urinary disorders) | 41 | 30
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Libido (Reproductive system and breast disorders) | 1 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 2 | 2
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 4 | 1
Vaginitis (Reproductive system and breast disorders) | 2 | 4
Vaginal Mucositis (Reproductive system and breast disorders) | 4 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 8 | 9
Syndromes - Other (General disorders) | 0 | 1
Flu-Like Syndrome (General disorders) | 1 | 2
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2014-04-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT00807768/Prot_000.pdf